CLINICAL TRIAL: NCT00560807
Title: Manual Therapy Dosage Factorial Study
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was stopped because the study never received funding
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Institutes of Health (NIH) (NIH); University of Western Ontario, Canada (Other)
Responsible Party: Joy MacDermid, McMaster University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1 R21 AT004263
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Whiplash Injuries
Keywords: WAD II; WAD III; mobilization; dosage; acute whiplash associated disorders (WAD) II and III (113) with a symptom duration of less than 30 days; neck pain
MeSH Terms: conditions — Whiplash Injuries; Weyers acrofacial dysostosis; Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (12):
- A (No Intervention): Zero treatment/3 weeks
- B (Active Comparator): Frequency of Mobilization:1/week Duration of Mobilization Treatment: 3 weeks
  Interventions: Procedure: Mobilization
- C (Active Comparator): Frequency of Mobilization: 1/week Duration of Mobilization Treatment: 6 weeks
  Interventions: Procedure: Mobilization
- D (Active Comparator): Frequency of Mobilization: 1/week Duration of Mobilization Treatment: 12 weeks
  Interventions: Procedure: Mobilization
- F (Active Comparator): Frequency of Mobilization: 2/week Duration of Mobilization Treatment: 3 weeks
  Interventions: Procedure: Mobilization
- G (Active Comparator): Frequency of Mobilization: 2/week Duration of Mobilization Treatment:6 weeks
  Interventions: Procedure: Mobilization
- H (Active Comparator): Frequency of Mobilization: 2/week Duration of Mobilization Treatment: 12 weeks
  Interventions: Procedure: Mobilization
- J (Active Comparator): Frequency of Mobilization: 3/week Duration of Mobilization Treatment: 3 weeks
  Interventions: Procedure: Mobilization
- K (Active Comparator): Frequency of Mobilization: 3/week Duration of Mobilization Treatment:6 weeks
  Interventions: Procedure: Mobilization
- L (Active Comparator): Frequency of Mobilization: 3/week Duration of Mobilization Treatment:12 weeks
  Interventions: Procedure: Mobilization
- E (No Intervention): Zero treatment/6 weeks
- I (No Intervention): Zero treatment/12 weeks

INTERVENTIONS:
Procedure: Mobilization — Mobilizations are passive movements performed in such a manner that the patient can volitionally prevent the movement. Types of mobilization include: a) passive oscillatory movements (2-3 Hz) of small or large amplitude, applied anywhere in a range of movement, typically for anything between 30 seconds and several minutes depending on the response and desired effects, and b) sustained stretching (glides) with or without tiny amplitude oscillations at the limit of the range.
  Arms: B; C; D; F; G; H; J; K; L

SUMMARY:
This study will determine biological responses to different dosages of neck mobilization intervention in patients, providing opportunities to identify the optimal dosage, predictors of response, outcome measures as well as the longitudinal changes in biology.

Subjects with acute whiplash associated disorders (WAD) II and III with a symptom duration of less than 30 days (acute) or 30 to 90 days (subacute) will be randomly assigned to receive different doses of mobilization. The dosage treatment groups will differ in the number of sessions (1, 2 or 3 times per week) and the duration of treatment (duration of treatment intervention will be 3, 6, or 12 weeks). A zero treatment/week option is included to insure that the impact of any mobilization is included and because previous studies suggest a single mobilization may have a treatment effect.

All patient participants will receive a core standard treatment of education, advice to stay active, and neck/postural stretching and strengthening exercise. All patient participants will receive supervised exercise and advice for the full 12 weeks. All patients will be provided with an instructional CD and exercise brochure to reinforce the whole program.

Follow-up assessments will consist of quantitative sensory testing (vibration threshold; current perception threshold), the Neck Walk Index (NWI), the Upper Cyclical Reach and Grasp Task, muscle biology analyses (cytokine analyses), central breathing control tests (capnography), range of motion, head flexion endurance, and self-report symptoms and disability (Visual Analogue Scale; Neck Disability Index; Disabilities of the Arm, Shoulder, Hand; pain threshold and tolerance algometry; and perceived self-efficacy; SF-36).

Hypothesis: During recovery, patient are expected to transition from an acute painful state to one where they can resume normal activity and add intensive strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* acute whiplash associated disorders (WAD) II and III (113) with a symptom duration of less than 30 days or subacute (30 to 90 days)
* pain in the neck but may radiate to the shoulder region or upper extremities or have an associated headache
* pain intensity must be at or above 30 mm on a 100 mm visual analogue scale
* must be a new episode of pain with ,no other occurrences of neck pain requiring treatment in the previous 4 months.

Exclusion Criteria:

* arthritis, neurological diseases, fractures, dislocation, rheumatoid arthritis, long tract signs and malignancy
* conditions that make the provision of neck exercise unsafe

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | Within 24 weeks
Current Perception Threshold (CPT) | Within 24 weeks
Neck Walk Index (NWI) | Within 24 weeks
Cyclical Reach and Grasp Test (CRGT) | Within 24 weeks
Muscle Biology (cytokine analyses) | Within 24 weeks
Central Breathing Control Test | Within 24 weeks
Neck Disability Index | Within 24 weeks
Pain Intensity - Visual Analogue Scale (VAS) | Within 24 weeks

SECONDARY OUTCOMES:
Global Perceived Effect (GPE) | Within 24 weeks
Disabilities of the Arm, Shoulder, and Hand (DASH) | Within 24 weeks
Pain Threshold and Pain Tolerance Algometry | Within 24 weeks
Head Flexion Endurance | Within 24 weeks
Range of Motion | Within 24 weeks
Quality of Life (SF-36v2) | within 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada